CLINICAL TRIAL: NCT06797414
Title: Comparison of Pilate Exercises With and Without Whole Body Vibration on Posture, Disability and Pain in Patient With Upper Cross Syndrome
Brief Title: Comparison of Pilate Exercises With and Without Whole Body Vibration in Patient With Upper Cross Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr Affifa
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Upper Cross Syndrome
Keywords: Whole Body Vibration; Rounded Shoulder Posture; Pilates Exercise; Upper Cross Syndrome; Young Adult
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: Will be treated with Pilate Exercises. Before applying exercise, hot pack will be applied for 15-20minutes.
  Interventions: Other: Pilate Exercises; Device: Hot Pack
- Group B (Active Comparator): Group B: Will be treated with WBV with Pilate Exercises. Before applying exercise, hot pack will be applied for 15-20minutes.
  Interventions: Other: Pilate Exercises; Other: Whole-body vibration; Device: Hot Pack

INTERVENTIONS:
Other: Pilate Exercises — PILATES EXERCISE METHODS:
  1. The cranium, triceps, back, and shoulder blades against the mat, then breath while maintaining muscle contraction .
  2. Arm circles (both directions) on the mat, then use strong ribcage breathing to connect into scapula.
  3. Diamond press: lie prone on a mat, using the lower part of the trapezius and serratusanterior muscles to slide shoulder blades out and down. Move into slight back extension maintaining this position.
  4. Diamond press: repeat above but add lateral arm movement to back extension .
  5. Arm slides 90°: lies supine on mat with arms bent at 90° and thumbs on floor. Slide elbows on floor toward waistline while contracting serratus anterior muscle.Repeat on the floor with other fingers. Always maintain proper neck alignment .
  6. Arm circles on a tiny barrel while lying on back with the head and neck supported by the barrel. Opened chest, then link the scapula to the barrel. Hold this position while performing arm circles.
Other: Whole-body vibration — Subjects were placed in a modified push-up position , put their hands in the middle of the platform, shoulder width apart, elbows slightly flexed, and their lower extremities were supported by kneeling on the floor . Vibration protocol included 5 sets of 60 s duration, at 5 mm amplitude and 30 Hz frequency, with a rest period of 60 s between sets . The subjects were reminded kneeling but upright and detached from the platform between sets.
  Arms: Group B
Device: Hot Pack — for 10 to 15 minutes

SUMMARY:
Nowadays, bad habits brought about by technology such as overuse of mobile phones, televisions, computers, and tablets, resulted in negative impacts on health. Bending in abnormal positions while using these devices causes various mechanical loads on the neck and upper back area, rounded shoulders from increased thoracic kyphosis etc., and this leads to poor posture that can cause UCS. Because of high prevalence of RSP especially in modern societies , proper treatment of this problem is necessary for prevention of further complications.There are different exercise regimes for RSP such as strengthening of lengthened muscles, scapular stabilizers, stretching of shorten muscles especially pectoral muscles, and soft tissue mobilization but Whole-Body Vibration (WBV) is a new method introduced since the last decade and there is no comparison available in the literature of upper cross syndrome between WBV with Pilate exercises on postural correction

The aim of the study is to compare effects Comparison of pilot exercises with and without whole body vibration on posture , disability and pain in patients with upper cross syndrome A randomized clinical trial will be conducted at PESSI.. Non-probability convenience sampling will be used, and 56 subjects, age 20-40 years will be randomly allocated into two groups by lottery method after meeting the inclusion criteria. Both groups will receive hot pack for 15-20 minutes and Pilate exercise perform both group as common treatment. Group A will be treated with pilate exercises and Group B will be treated with pilate exercise with whole body vibration Both groups received two sessions per week for four consecutive weeks by another well trained physical therapist. Session duration for both groups ranged from 55 minutes to 1 hour. 2 sessions per week and total 8 sessions for 4 weeks. The outcome measures will be conducted through NPRS,NDI,RSP WAS MEASURED IN SUPINE POSITION AND THEN PML AND TSD before and after 4 weeks. Data will be analyzed using SPSS software version 26.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rounded shoulder
* Forward head
* Having a moderate level of physical activity
* RSP measurement in supine n>1 inch(12)
* NPRS >3(18)
* NDI > 10(19)

Exclusion Criteria:

* Pregnant, having untreated wounds, joint or artificial limb
* Suffering from diseases such as-malignancy, diabetes, epilepsy, acute thrombosis, acute migraine, acute infectious conditions, and tumor having history of neurological diseases like vestibulr disease, stroke, kidney or bladder stones, and finally reporting history of back problems such as herniated disk and deformities like scoliosis. experienced any recent trauma (within three months of the initial consultation)
* Chief complaint of headaches or facial pain , hypertension, osteoporosis, and presence of any structural abnormality in the upper and middle back (e.g., scoliosis or presence of positive Adam's test) .
* Participants on anti-inflammatory or muscle relaxant medications were given a three-day period "wash out" before participating in the study (13).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-02-07 (Estimated); Study Completion 2025-02-07 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | baseline, after 4 weeks
  Numeric Pain Rating Scale (NRS-11), which is an eleven-point scale in which the end points are the extremes of no pain at all (score of 0) and the worst pain the patient has ever experienced (score of 10). NPRS-11 pain severity score of "4" is frequently given special significance in this regard, suggesting it as a potential threshold value for pain severity in clinical practice(20).
  scale has high reliability (0.95-0.96)(21).
NDI for neck disability (Urdu version) | baseline, after 4 weeks
  In 1991, Howard Vernon developed the Neck Disability Index (NDI)(22). The Neck Disability Index (NDI) was the first tool to measure self-reported disability in patients with neck pain. It is used extensively in literature and its psychometric properties have been well established. It has been translated and cross-culturally adapted to many languages. The index has 10 neck-related functional activities scored on a 0-5 scale for each item and a total raw score of 50. The higher the score, the greater the disability(23).
  NDI-U is a reliable, valid and responsive questionnaire to measure disability in Urdu- speaking patients with CMNP(24).

SECONDARY OUTCOMES:
Rounded Shoulder Posture Was Measured In Supine Position And Then Pml And Tsd ( By measuring tape manually) | baseline, after 4 weeks
  Supine measurement of RSP:
  Iis the distance between the posterior aspect of the lateral acromion process and the exam table in the supine position . An investigator marks the posterior aspect of the lateral acromion process while the subject is in the supine position, with the shoulder in neutral position to avoid measurement variations due to humeral rotation . The investigator then measures the distance from the table to the posterior aspect of the lateral acromion process by using a straight ruler and records the value in inches
  PML:
  Is the distance from the inferomedial aspect of the coracoid process to the caudal edge of the fourth rib at the sternum . The investigator marks the distance between the inferomedial aspect of the coracoid process and the caudal edge of the fourth rib at the sternum while the subject stands in a relaxed position then records the distanc between the two marked points in inches with a tapeline .

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, MS, Principal Investigator — Riphah International University
Locations (1):
- Punjab Employees Social Security Institution, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No